CLINICAL TRIAL: NCT00807430
Title: A Single Centre, Randomised, Clinical Placebo Controlled Study of the Optimal Treatment and Long-term Effect of FES on Bruxism
Brief Title: Treatment Period and Long-term Effect of Functional Electric Stimulation (FES) for Bruxism
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Medotech A/S (Industry)
Responsible Party: Peter Svensson, Aarhus University Dentist School
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMD-00
Record Dates: First submitted 2008-12-09; First posted 2008-12-11 (Estimated); Last update posted 2009-10-21 (Estimated); Status verified 2009-10

CONDITIONS: Bruxism
Keywords: Bruxism; EMG; Biofeedback
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 24 patients receiving active treatment
  Interventions: Device: Grindcare (Active)
- 2 (Placebo Comparator): Placebo treatment
  Interventions: Device: Grindcare (Placebo - the device is not activated)

INTERVENTIONS:
Device: Grindcare (Active) — Active treatment
  Arms: 1
Device: Grindcare (Placebo - the device is not activated) — Placebo treatment
  Arms: 2

SUMMARY:
To investigate the effect of the treatment with Grindcare® on the muscles- and jaw symptoms and at the jaw muscle activity during sleep.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated ICF
* 18 years or older
* Fulfill the RDC-criteria for myofascial TMD diagnose (group 1a or 1b)
* Average pain more that 3 on a Visual Analog scale (VAS) in the baseline period

Exclusion Criteria:

* Contraindication of concommitant diseases for the study judged by investigator
* Daily use of pain medication, e.g. prophylaxis against migraine or headache.
* Patients who are using occlusal splints in the treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Primary outcome is to reduce the EMG activity per hour per night | 10 weeks after start of treatment

SECONDARY OUTCOMES:
Secondary outcome is to evaluate long-term effect of FES om EMG activity | after end of treatment with FES

CONTACTS AND LOCATIONS:
Overall Officials: Troels B Mortensen, Study Director — Medotech A/S
Locations (1):
- Odontologisk Institut, Aarhus C, Denmark